CLINICAL TRIAL: NCT01582516
Title: A Phase I/II Trial of a Conditionally Replication-competent Adenovirus (Delta-24-rgd) Administered by Convection Enhanced Delivery in Patients With Recurrent Glioblastoma
Brief Title: Safety Study of Replication-competent Adenovirus (Delta-24-rgd) in Patients With Recurrent Glioblastoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, C.Dirven, MD PhD, Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL24958.000.08
Record Dates: First submitted 2012-04-19; First posted 2012-04-20 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2015-03

CONDITIONS: Brain Tumor; Recurring Glioblastoma
Keywords: brain tumor; virotherapy; glioblastoma; replication competent adenovirus
MeSH Terms: conditions — Brain Neoplasms; Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Delta24-RGD (Experimental): Intracerebral slow continuous infusion of study drug in increasing dose
  Interventions: Biological: delta-24-RGD adenovirus

INTERVENTIONS:
Biological: delta-24-RGD adenovirus — slow continuous microinfusion in and around the brain tumor during 44 hrs.by 4 temporary placed catheters

SUMMARY:
In the Netherlands a 2 center investigator-driven phase I/II clinical trial is initiated in June 2010 testing the oncolytic adenovirus Delta24-RGD to treat glioblastoma patients. The virus is administrated using convection-enhanced delivery by 4 catheters as delivery technique, targeting solid tumor as well as infiltrated tumor cells within the peri-tumoral brain. Patients will be enrolled in cohorts of 3 per dose-level. The dose levels to be explored are: 10^7, 10^8, 10^9, 10^10, 3*10^10 and 10^11 viral particles (vp). Once the MTD has been determined, or the study has reached the highest dose cohort, a further 6 or 9 patients will be enrolled at the MTD and evaluated for safety and preliminary signs of efficacy, such that in total at least 12 patients have received the MTD.

The primary objective is to determine the safety and tolerability of Delta-24-RGD administered by CED to the tumor and the surrounding infiltrated brain in patients with recurrent GBM. Secondary objectives are to determine the Progression Free Survival (PFS), Overall Survival (OS), and tumor response rate in patients with recurring tumors amenable for surgical resection and treated at the MTD.

Cerebrospinal fluid as well as brain interstitial fluid by microdialysis next to the routinely collected samples of blood at various timepoints before, during and after virus infusion. Various neurodegenerative biomarkers as well as markers of immune response will be assessed in these samples.

Furthermore extensive sampling and PCR analyses will be performed to evaluate distribution and shedding of the virus.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically proven primary Glioblastoma Multiforme (GBM) will be eligible for this protocol.
2. Patients must show unequivocal evidence for tumor recurrence or progression by MRI scan within 3 weeks prior to registration after failing prior resection (surgery or biopsy) and/ or chemo- and/or radiation therapy.
3. Recurring tumors must either be accessible for surgery, or , when not accessible for surgery meet the following criteria:

   1. unifocal
   2. midline shift < 0.5 cm
   3. no radiological signs of uncal herniation
4. All recurring tumors must be restricted to one hemisphere, without signs of subependymal spreading.
5. Before start of virus treatment histological analysis of the resected, or biopsied tumor recurrence must confirm the diagnosis of GBM (based on frozen section).
6. Patients may or may not have had prior chemotherapy.
7. Patients must be able to read and understand the informed consent document and must sign and date the informed consent. Procedures to obtain such informed consent should be according to ICH-GCP, the local regulatory requirement and the rules followed at the institute.
8. Patients must be > 18 and < 75 years old.
9. Patients must have a Karnofsky performance status rating > 70 (Appendix 2).
10. Patients must have recovered from the toxic effects of prior therapy. For example, they must be at least two weeks after vincristine, 6 weeks after nitrosoureas, 3 weeks after procarbazine or temozolomide administration, and 6 weeks after radiation therapy.
11. If sexually active, patients must be willing to use barrier contraception for the duration of the study.
12. Patients must have adequate hepatic, renal and bone marrow function, defined as

    * absolute neutrophil count (ANC) > 1,5* 109/L
    * platelet count of > 100* 109/L
    * ALT (SGPT), AST (SGOT) and Alkaline Phosphatase < 2 times ULN
    * total bilirubin <1.5 mg/dL
    * creatinine <1.5 times ULN
    * urea (BUN) <1.5 times ULN

Exclusion Criteria:

1. Patients with active uncontrolled infection. Upper pulmonary infection and flu-like signs or presence of adenovirus in pre-operative throat-swab or serum sample as determined by PCR. All patients must be afebrile (<38.0 C) at the start of therapy
2. Evidence of bleeding diathesis or use of anticoagulant medication.
3. Patients with systemic diseases or other unstable conditions which may be associated with unacceptable anesthetic/ operative risk and/or which would not allow safe completion of this study protocol, e.g. uncontrolled seizures.
4. Because of the potential risk of a recombinant virus containing a gene involved in cellular growth regulation and differentiation which could potentially affect a developing fetus or growing infant, females who are pregnant, at risk of pregnancy, or breast feeding a baby during the study period are excluded.
5. Because of the potential risk of serious infection in immune-compromised individuals, patients known to have HIV infection are excluded.
6. Patients with a known germline deficit in the retinoblastoma gene or its related pathways.
7. Patients with other primary malignancy than GBM. However, patients with curatively treated carcinoma-in situ or basal cell carcinoma or patients who have been disease free for at least 2 years and not using any anti-cancer therapy, are eligible.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
treatment related serious adverse events | untill 3 months after treatment

SECONDARY OUTCOMES:
The number of participants alive after 6 months and after 1 year : Progression free survival after 6 months and overall survival after 6 months and one year. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Clemens Dirven, MD PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- ERasmus Medical Center, Rotterdam, Netherlands